CLINICAL TRIAL: NCT06620458
Title: A Retrospective Study on the Factors of Drug-coated Balloon Restenosis
Acronym: RE-DCB
Status: Recruiting | Type: Observational
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Other Study IDs: HenanICE202403
Record Dates: First submitted 2024-04-28; First posted 2024-10-01 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
Keywords: DCB CHD IVUS OCT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to analyze potential factors post paclitaxel drug-coated balloon angioplasty in patients with Denovo large vessels disease. It includes imaging endpoints and clinical event endpoints. Over 5000 patients are expected to be enrolled.

DETAILED DESCRIPTION:
This study is a retrospective analysis that retrospectively reviewed over approximately 5000 patients with de novo-large-vessel disease who underwent paclitaxel drug-coated balloon angioplasty. The study endpoints include cardiovascular adverse events at 1 year (cardiovascular death, cardiovascular events) and coronary angiographic outcomes (primarily late lumen loss, restenosis rate). It primarily focuses on differences in baseline characteristics, lesion features, intracavitary imaging characteristics(Including OCT, IVUS), hemodynamic parameter，and procedural approaches among patients. Over 5000 patients are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age:

  18 years and older.
* Diagnosis:

Diagnosed with coronary artery disease with native large vessel lesions confirmed by coronary angiography.

* Treatment Plan:

Scheduled to receive paclitaxel drug-coated balloon angioplasty.

* Informed Consent:

Patients have been fully informed about the nature and purpose of the study, and have voluntarily agreed to participate, with signed informed consent.

* Physiological Status:

Cardiac function classified as NYHA I-III.

Exclusion Criteria:

* Allergy History:

Known allergies to paclitaxel or any materials used in angioplasty (e.g., contrast agents).

* Severe Complications:

Uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg).

* Other Medical Conditions:

Active bleeding or clotting disorders.

* Other serious diseases with a life expectancy of less than 1 year (e.g., advanced cancer).
* Pregnancy or Nursing: Women who are currently pregnant or breastfeeding.
* Participation in Other Studies: Currently participating in other clinical trials that might affect the results of this study.
* Psychological or Behavioral Factors: History of psychiatric or behavioral disorders that could interfere with adherence to study protocols, or communication barriers that prevent understanding of study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study targets adults aged 18 and over who have been diagnosed with coronary artery disease featuring native large vessel lesions and are scheduled to undergo paclitaxel drug-coated balloon angioplasty.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
MACE | 12 months
  cardiovascular adverse events:defined as death, Myocardial Infarction (MI, Q waves and non-Q waves), emergent cardiac bypass surgery, or any target lesion revascularization (repeat Percutaneous transluminal coronary angioplasty (PTCA) or Coronary artery bypass grafting (CABG)).

SECONDARY OUTCOMES:
LLL(late lumen loss) | 12 months
  Detection by QCA technique by subtracting the minimum lumen diameter at review from the minimum lumen diameter in the immediate postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, Ph.D, Study Chair — Fuwai central China cardiovascular hospotial
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, China